CLINICAL TRIAL: NCT03753529
Title: Effect of Manual Therapy on Jaw Movement and Function in Patients With Bruxism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, HAhmed, lecture of biomechanics, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/001936
Record Dates: First submitted 2018-11-02; First posted 2018-11-27 (Actual); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: Bruxism; TMJ Pain
MeSH Terms: conditions — Bruxism | interventions — Continuous Positive Airway Pressure; Acupressure; Control Groups; Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- deep friction massage group (Experimental)
  Interventions: Other: Deep friction massage
- pressure release group (Experimental)
  Interventions: Other: Pressure release
- control group (Experimental)
  Interventions: Other: control group

INTERVENTIONS:
Other: Deep friction massage — Submitted to three session weekly 30-minute sessions of therapy will performed by the administration of sliding and kneading maneuvers of the masseter and temporalis muscles, bilaterally,lateral pterygoid and digastric over four consecutive weeks (total:12 sessions) Sliding consisted of a unidirectional movement in which part of the therapist's hand (mainly the fingertips) will used, moving from the proximal to the distal portion of the face with constant, progressive pressure compatible with the status of each tissue. The degree of pressure varied depending on the level of pain, sensitivity and tension in each individual. Kneading consisted of a gripping maneuver of a muscle group or portion of a muscle.Then follow-up with a passive stretch to the muscle. This will repeated for three to five times for three sessions per week for 4 weeks.
  Arms: deep friction massage group
Other: Pressure release — First, using a pincer grasp moved throughout the fibers of the pterygoid, masseter, digastric and temporalis muscles to palpate the muscle aiming to locate a trigger point . A common location is detected according to Simon and Travell book. Once located on the trigger point, apply an IC by gradually applying pressure to the trigger point with your thumb. Keep in communication with the patient, checking to ensure that in staying within the limits of his pain tolerance. Hold this technique for approximately 20 seconds to 1 minute, patient tells you that pain has diminished, or until feels the muscle fibers begin to relax under your pressure. Once feel this release, gradually release pressure. All identified trigger points were treated. Then follow-up with a passive stretch to the muscle. This will repeated for three to five times for three sessions per week for 4 weeks.
  Other Names: Ischemic pressure and ischemic compression (IC)
  Arms: pressure release group
Other: control group — Stretching and transcutaneous electrical nerve stimulation
  Other Names: Stretching and transcutaneous electrical nerve stimulation
  Arms: control group

SUMMARY:
Hypothesis

1. There will be no significant statistical effect of Trigger Point Pressure release and Deep striking massage on pain level in patients with bruxism.
2. There will be no significant statistical effect of Trigger Point Pressure release and Deep striking massage on Range of Motion in patients with bruxism.
3. There will be no significant statistical effect of Trigger Point Pressure release and Deep striking massage on Sleep Quality Index in patients with bruxism.
4. There will be no significant statistical effect of Trigger Point Pressure release and Deep striking massage on proprioception awareness in patients with bruxism.
5. There will be no significant statistical effect of Trigger Point Pressure release and Deep striking massage on Stress in patients with bruxism.
6. There will be no significant statistical effect of Trigger Point Pressure release and Deep striking massage on Anxiety in patients with bruxism.
7. There will be no significant statistical effect of Trigger Point Pressure release and Deep striking massage on Temporomandibular (TMJ) function in patients with bruxism.
8. There will be no significant statistical effect of Trigger Point Pressure release and Deep striking massage on Oral Health Impact Profile in patients with bruxism.

ELIGIBILITY:
Inclusion Criteria:

1. The volunteers diagnosed with bruxism based on the criteria of the American Academy of Sleep Medicine
2. Positive self-report of awake bruxism.
3. Self-report of muscle fatigue or tenderness on awakening.
4. Sleeping partner reports of grinding sounds during the night in the last 6 months, or awake clenching.

Exclusion Criteria:

1. Severe psychological disorder and/or the use of antipsychotic psychotropic drugs(with the exception of anxiety and depression).
2. Using medications that influence sleep or motor behavior.
3. Direct trauma or past surgery in the orofacial region.
4. On physical, speech, dental, or psychological therapy at the time of study entry.
5. Currently undergoing physical therapy for TMD.
6. Neurological or central nervous system and/or peripheral nervous system disorders or history of neuromuscular disease.
7. The presence of prosthesis or extensive prosthetic restorations and the presence of gross malocclusion.
8. More than two missing teeth, except third molars;
9. Systemic and/or degenerative diseases.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2020-01 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
changes of Trigger point pressure pain threshold | Pre- and post-treatment (twelve treatment sessions within one month, three sessions per week).
  To compare pressure pain threshold (PPT) values for selected muscles (temporalis, masseter, digastric and lateral pterygoid) in patients with bruxism before and after treatment using Pressure Algometer.
Changes of mandibular range of motion at month of treatment | Pre- and post-treatment (twelve treatment sessions within one month, three sessions per week).
  Vernier caliper used to measure opening, lateral movements, protraction and retraction.

SECONDARY OUTCOMES:
Changes of proprioception awareness | Pre- and post-treatment (twelve treatment sessions within one month, three sessions per week).
  Measure ability of patient before treatment and after to move mandible to specific angle(measured by vernier caliper) identified before test
Stress | Pre- and post-treatment (twelve treatment sessions within one month, three sessions per week).
  Using Perceived Stress Scale to measure stress which consist of 10 items. The 10 items in the scale inquire about feelings and thoughts that tap the degree to which respondents find their current life situation unpredictable, uncontrollable and stressful. Respondents indicate how often in the past month they have felt or thought a certain way on a 5-point Likert scale (0 = never, 1 = almost never, 2 = sometimes, 3 = fairly often, 4 = very often). The higher the score the higher the perceived stress is. The scale correlates with different psychosocial measures specifically depression, anxiety, and perception of poor health as well as with decreased satisfaction with self, job and life in general.
Anxiety | Pre- and post-treatment (twelve treatment sessions within one month, three sessions per week).
  Measured using the State-triat Anxiety Inventory. It consists of two independent scales, with 20 questions each, measuring anxiety as a trait (in general) and as a state (at the moment). Each question is scored (from 1 to 4), and scores for the scales range from 20 to 80 as follows: mild anxiety (20 to 34); moderate anxiety (35 to 49); high anxiety (50 to 64); and very high anxiety (65 to 80).
Changes of quality of sleep at month of treatment | Pre- and post-treatment (twelve treatment sessions within one month, three sessions per week).
  Using The Pittsburgh Sleep Quality Index, It consists of 19 questions grouped under seven domains: subjective sleep quality; sleep latency; sleep duration; usual sleep efficiency; sleep disturbances; use of medications; and diurnal dysfunction. Each domain is scored (0 to 3) and a total score (0 to 21) is calculated as follows: scores ranging from 0 to 4 are indicative of good sleep quality; scores from 5 to 10 suggest poor sleep quality; scores above 10 are suggestive of sleep disorders. Five other questions are answered by participants' spouses or partners, and further characterize sleep quality.
Temporomandibular (TMJ) function | Pre- and post-treatment (twelve treatment sessions within one month, three sessions per week).
  Using Temporomandibular Disorder (TMD) Disability Index Questionnaire,The TMD Disability Index consists of ten questions regarding disability associated with TMD, and each question is scored from 0-4. Higher scores represent greater levels of disability.
Changes in Oral Health Impact Profile. | Pre- and post-treatment (twelve treatment sessions within one month, three sessions per week).
  using Oral Health Impact Profile.(OHIP), The OHIP-14 is a 14-items questionnaire designed to measure self-reported functional limitation that focuses on seven dimensions of impact (functional limitation, pain, psychological discomfort, physical disability, psychological disability, social disability and handicap) with participants being asked to respond according to frequency of impact on a 5-point Likert scale coded never (score 0), hardly ever (score 1), occasionally (score 2), fairly often (score 3) and very often (score 4) using a twelve-months recall period.